CLINICAL TRIAL: NCT03441087
Title: Ultrasound and Hysteroscopy's Place on the Diagnosis of Abnormal Uterin Bleeding
Brief Title: The Role of TVSG and HS in Determining Endometrial Pathologies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Nazlı YENIGUL, Principal Investigator MD, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 349
Record Dates: First submitted 2018-02-15; First posted 2018-02-22 (Actual); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Abnormal Uterine Bleeding
Keywords: transvaginal ultrasonography; hysteroscopy; abnormal uterine bleeding
MeSH Terms: conditions — Metrorrhagia | interventions — Hysteroscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transvaginal ultrasound (Other): Transvaginal ultrasound was applied 216 women with abnormal uterine bleeding.The transvaginal ultrasound diagnoses were compared with the received endometrial samples.
  Interventions: Device: Transvaginal ultrasound
- Hysteroscopy (Other): Hysteroscopy was also performed under general anesthesia.Hysteroscopy was performed by a single operator (NNY).The operator and two supervising endoscopists were blinded to the ultrasound results.After the hysteroscopy, endometrial sampling was also done. The diagnoses were compared with the received endometrial samples.
  Interventions: Device: Hysteroscopy

INTERVENTIONS:
Device: Transvaginal ultrasound
  Arms: Transvaginal ultrasound
Device: Hysteroscopy
  Arms: Hysteroscopy

SUMMARY:
Although hysteroscopy (HS) and transvaginal ultrasonography (TVSG) are methods in the diagnosis of AUB, there is some suspicion about their efficacy. The aim of this study was to determine the efficacy and safety of HS and TVSG on diagnosing abnormal uterine bleeding(AUB) .216 women admitted to the investigators clinic (Sisli Ethal Training and Research Hospital, Obstetrics and Gynecology Department Obstetrics Service ) between 21-51 years of age. These patients were divided into two groups; menopause (71women) and pre-menopause (145 women). HS and endometrial sampling were performed both groups after TVSG.The success of these methods was assessed by kappa analysis

ELIGIBILITY:
Inclusion Criteria:

* patients who have no history of hysteroscopy and curettage,
* patients who have no history of ovulatory dysfunction
* women who have active vaginal bleeding.

Exclusion Criteria:

* presence of genital infections/PID
* presence of pregnancy
* presence of vaginal or cervical pathology causing vaginal bleeding
* women who are receiving hormonal treatment (COC/HRT)
* patients formerly diagnosed with endometrial pathology
* patients having coagulopathy
* women who are using intrauterine device.

Ages: 21 Years to 51 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 216 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2011-12-31 (Actual); Study Completion 2011-12-31 (Actual)

PRIMARY OUTCOMES:
accuracy of diagnostic performance transvaginal ultrasonography and hysteroscopy | up to 12 month
  The main outcome variable of the study was accuracy of diagnostic performance of transvaginal ultrasonography and hysteroscopy in premenopausal and menopausal women with abnormal uterin bleeding .

CONTACTS AND LOCATIONS:
Overall Officials: Nefise Nazlı YENIGUL, MD, Study Director — Sisli Etfal Research and Training hospital, Obstetrics and gynecology department Istanbul, Marmara Turkey